CLINICAL TRIAL: NCT00515671
Title: Illness Management and Recovery for Veterans With Severe Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Indiana University (Other); Dartmouth College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IAC 05-254
Record Dates: First submitted 2007-08-10; First posted 2007-08-14 (Estimated); Results first posted 2014-10-10 (Estimated); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Schizophrenia; Schizo-affective Disorder
Keywords: self-management; recovery; severe mental illness
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders | interventions — Salvage Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1_IMR (Experimental): Illness Management and Recovery was offered in small groups (less than 8), co-facilitated by either an experienced masters level clinician or a doctoral level psychologist and by a doctoral student in clinical psychology. Facilitators used the IMR curriculum, incorporating psychoeducation, cognitive-behavioral approaches, relapse prevention, social skills training, and coping skills training. Facilitators worked with groups to set personal recovery goals and address progress towards those goals throughout the intervention. Home assignments helped participants apply newly learned skills and/or make progress on goals. Groups were open to rolling admission across the study period
  Interventions: Behavioral: Illness Management and Recovery
- Arm 2_PS (Placebo Comparator): Problem Solving was the active control condition (also offered in groups weekly for 9 months). Participants were encouraged to discuss current concerns and receive group support; we did not use structured problem solving tasks. These groups were led by the same facilitators described above, who helped establish group expectations (attendance, confidentiality), encouraged participation, and provided process-oriented observations; there was no formal curriculum, goal setting, or homework assignments.
  Interventions: Behavioral: Problem Solving

INTERVENTIONS:
Behavioral: Illness Management and Recovery — a structured curriculum to help mental health consumers manage their illnesses and pursue goals related to recovery from mental illness
  Other Names: IMR
  Arms: Arm 1_IMR
Behavioral: Problem Solving — Weekly problem-solving support group
  Other Names: PS
  Arms: Arm 2_PS

SUMMARY:
The President's New Freedom Commission on Mental Health has called for a transformation of the mental health system to partner with consumers of those services in delivering effective interventions focused on recovery, and the Department of Veterans Affairs (VA) has developed a Mental Health Strategic Plan to address these recommendations. One promising approach is to implement Illness Management and Recovery (IMR), a structured curriculum to help mental health consumers manage their illnesses and pursue goals related to recovery from mental illness.

IMR was developed from a review of effective approaches for illness self-management training in persons with severe mental illness. The 9-month curriculum is taught using motivational, educational, and cognitive-behavioral techniques, and incorporates five evidence-based practices: education about mental illness, strategies for increasing medication adherence, skills training to enhance social support, relapse prevention planning, and coping skills training. The program was developed for widespread dissemination and includes a manual, worksheets, an introductory video, a clinical training video, a fidelity scale, and informational brochures for consumers, family members, clinicians, and administrators.

DETAILED DESCRIPTION:
Background:

The President's New Freedom Commission on Mental Health has called for a transformation of the mental health system to partner with consumers of those services in delivering effective interventions focused on recovery, and the Department of Veterans Affairs (VA) has developed aMental Health Strategic Plan to address these recommendations. One promising approach is to implement Illness Management and Recovery (IMR), a structured curriculum to help mental health consumers manage their illnesses and pursue goals related to recovery from mental illness.

IMR was developed from a review of effective approaches for illness self-management training in persons with severe mental illness. The 9-month curriculum is taught using educational, motivational, and cognitive-behavioral techniques, and incorporates five evidence-based practices: education about mental illness, strategies for increasing medication adherence, skills training to enhance social support, relapse prevention planning, and coping skills training. The program was developed for widespread dissemination and includes a manual, worksheets, an introductory video, a clinical training video, a fidelity scale, and informational brochures for consumers, family members, clinicians, and administrators.

Objective:

Although IMR is based on practices shown to be effective in controlled research, effectiveness of the comprehensive package of IMR has not yet been demonstrated in a randomized, controlled trial. The primary aim of the proposed research is to test the effectiveness of IMR as an implementation package. Our primary focus is to examine the impact of IMR intervention on consumer outcomes related to illness self-management and recovery.

Methods:

This is a randomized, controlled trial comparing IMR to usual mental health treatment, with an attention-control group in 200 veterans with schizophrenia spectrum disorders. Assessment will include semi-structured interviews and standardized measures at baseline, 9 months, and 18 months to assess illness self-management (e.g., symptoms), objective indicators of recovery (e.g., role functioning), and subjective indicators of recovery (e.g., perceptions of well-being). Electronic medical records will be accessed to determine the impact of IMR on other service utilization and costs.

Impact:

The proposed study directly addresses a stated need in the VA's Mental Health Strategic Plan and is a critical first step to systematically evaluating the effectiveness of a comprehensive, manual-based approach to improving recovery outcomes for veterans with severe mental illness. As an implementation package, IMR offers mental health providers useful tools that could be widely disseminated across the VA system.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving (or newly admitted to) mental health services from any mental health treatment programs at the Roudebush VAMC or Midtown Community Mental Health Center (MCMHC) in Indianapolis, IN
* Age 18 or older
* SCID-confirmed diagnosis of schizophrenia or schizoaffective disorder
* Stated interest in learning more about their illness
* Willing and able to give informed consent

Exclusion Criteria:

* Severe medical condition that would limit participation in an 18-month study (e.g., end stage renal disease, metastatic cancer, life expectancy less than 18 months; if participant is unsure, with permission will contact primary physician)
* Evidence of dementia or severe cognitive dysfunction on cognitive screener

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2008-01; Primary Completion 2012-04 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle P Salyers, MS PhD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Frankel RM, Salyers MP, Bonfils KA, Oles SK, Matthias MS. Agenda setting in psychiatric consultations: an exploratory study. Psychiatr Rehabil J. 2013 Sep;36(3):195-201. doi: 10.1037/prj0000004. Epub 2013 Jul 1. PMID 23815174
- [Result] McGuire AB, Bonfils KA, Kukla M, Myers L, Salyers MP. Measuring participation in an evidence-based practice: illness management and recovery group attendance. Psychiatry Res. 2013 Dec 30;210(3):684-9. doi: 10.1016/j.psychres.2013.08.008. Epub 2013 Sep 5. PMID 24011850
- [Result] Matthias MS, Salyers MP, Frankel RM. Re-thinking shared decision-making: context matters. Patient Educ Couns. 2013 May;91(2):176-9. doi: 10.1016/j.pec.2013.01.006. Epub 2013 Feb 11. PMID 23410979
- [Result] McGuire AB, Kukla M, Green A, Gilbride D, Mueser KT, Salyers MP. Illness management and recovery: a review of the literature. Psychiatr Serv. 2014 Feb 1;65(2):171-9. doi: 10.1176/appi.ps.201200274. PMID 24178191
- [Result] Salyers MP, McGuire AB, Kukla M, Fukui S, Lysaker PH, Mueser KT. A randomized controlled trial of illness management and recovery with an active control group. Psychiatr Serv. 2014 Aug 1;65(8):1005-11. doi: 10.1176/appi.ps.201300354. PMID 24733680
- [Result] McGuire AB, Stull LG, Mueser KT, Santos M, Mook A, Rose N, Tunze C, White LM, Salyers MP. Development and reliability of a measure of clinician competence in providing illness management and recovery. Psychiatr Serv. 2012 Aug;63(8):772-8. doi: 10.1176/appi.ps.201100144. PMID 22854724
- [Result] Tsai J, Salyers MP, McGuire AB. A cross-sectional study of recovery training and staff attitudes in four community mental health centers. Psychiatr Rehabil J. 2011 Winter;34(3):186-93. doi: 10.2975/34.3.2011.186.193. PMID 21208857

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Receives IMR groups once a week for 9 months in addition to care as usual.
  Illness Management and Recovery Training: a structured curriculum to help mental health consumers manage their illnesses and pursue goals related to recovery from mental illness
- Arm 2: Receives support groups once a week for 9 months in addition to care as usual.
  Illness Management and Recovery Training: a structured curriculum to help mental health consumers manage their illnesses and pursue goals related to recovery from mental illness
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 60 | 58
Completed | 43 | 41
Not Completed | 17 | 17
Not completed — Lost to Follow-up | 13 | 10
Not completed — Withdrawal by Subject | 3 | 5
Not completed — incarcerated | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 60 | 58 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (9.3) | 47.6 (8.5) | 47.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 46 | 48 | 94
Race/Ethnicity, Customized [Number; unit: participants]
  white | 22 | 18 | 40
  African American | 32 | 40 | 72
  More than one | 6 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 60 | 58 | 118

OUTCOME MEASURES:

1. Primary Outcome: Illness Management Ratings
Description: Illness self-management was assessed with the consumer-rated Illness Management and Recovery Scale. Items are rated on a 5-point behaviorally anchored scale; the mean across all 15 items forms an overall score of illness management (ranging from 1 to 5), with higher scores indicating better self-management.
Time Frame: Baseline, 9 months, 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 60 | 58
units on a scale
  Illness Management-baseline | 3.5 (.5) | 3.3 (.5)
  Illness Management-9 months | 3.5 (.6) | 3.6 (.6)
  Illness Management - 18 months | 3.6 (.5) | 3.5 (.6)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p = .8868, Mixed Models Analysis

2. Secondary Outcome: Psychiatric Symptoms (PANSS Total)
Description: Psychiatric symptomatology was assessed by the Positive and Negative Syndrome Scale (PANSS), a widely-used, 30-item rating scale. The PANSS has previously demonstrated satisfactory internal consistency, test-retest reliability, and validity. Raters were trained to reach inter-rater agreement of .80 prior to interviewing participants. This is the total score, which ranges from 30 to 210, with higher scores indicating more severe symptoms.
Time Frame: Baseline, 9 months, 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 60 | 58
units on a scale
  Total Symptoms - Baseline | 75.1 (16.1) | 76.1 (15.3)
  Total Symptoms - 9 months | 68.5 (18.5) | 66.6 (14.9)
  Total Symptoms - 18 months | 61.9 (17.1) | 65.3 (19.6)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p = .3328, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/58
Other Adverse Events (participants affected / at risk) | 0/60 | 0/58

LIMITATIONS AND CAVEATS:
Low attendance in both groups, may not have had enough "exposure" Study embedded in a treatment-rich environment, cannot sort out other impacts on outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No